CLINICAL TRIAL: NCT01748552
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Oral Doses of LY2922083 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2922083 in Healthy Participants and Participants With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14793; I6J-FW-PRBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2922083

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Part A) (Placebo Comparator): Single oral dose of placebo administered to healthy participants in up to 1 of 3 study periods in Part A
  Interventions: Drug: Placebo
- LY2922083 (Part A) (Experimental): Single ascending dose of LY2922083 (starting at 0.5 milligrams [mg]) administered orally to healthy participants in up to 2 of 3 study periods in Part A
  Interventions: Drug: LY2922083
- Placebo (Part B) (Placebo Comparator): Single oral dose of placebo administered to participants with type 2 diabetes mellitus (T2DM) in up to 1 of 3 study periods in Part B
  Interventions: Drug: Placebo
- LY2922083 (Part B) (Experimental): Single ascending dose of LY2922083 administered orally to participants with T2DM in up to 2 of 3 study periods in Part B. Dose determined by Part A
  Interventions: Drug: LY2922083

INTERVENTIONS:
Drug: Placebo — Administered orally as capsules
  Arms: Placebo (Part A); Placebo (Part B)
Drug: LY2922083 — Administered orally as capsules
  Arms: LY2922083 (Part A); LY2922083 (Part B)

SUMMARY:
The aim of this trial is to evaluate the safety of the study drug in healthy participants and participants with diabetes. It will investigate how much of the study drug gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected.

The study consists of two parts. Part A will study healthy participants in up to 3 dosing periods over approximately 6 weeks. Part B will study participants with diabetes in up to 3 dosing periods over approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

For all participants :

* Must be a male, or a female who cannot become pregnant, and who is either a healthy participant, or who has type 2 diabetes
* Have a screening body mass index (BMI) of at least 18.0 kilograms per square meter (kg/m^2)
* Have blood pressure, pulse rate, blood and urine laboratory test results acceptable for the study

For participants with T2DM:

* Do not have any change to their diabetes treatment (exercise with or without metformin) for at least 4 weeks prior to screening
* Have a glycated hemoglobin (HbA1c) value of greater than or equal to 6% and less than or equal to 11% at screening

Exclusion Criteria:

For all participants :

* Are currently participating in another clinical study or completed one in the last 30 days
* Are allergic to LY2922083 or other related drugs
* Have a history of significant heart, lung, liver, kidney, stomach or brain disease, or have any medical problems which may cause an increased risk during the study
* Have electrocardiogram (ECG) readings that are not suitable for the study
* Have a history of hepatitis or jaundice
* Are infected with hepatitis B
* Are infected with hepatitis C
* Are infected with human immunodeficiency virus (HIV)
* Have donated more than 450 milliliters (mL) of blood in the last 3 months or have donated any blood in the last month
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female), or are unwilling to stop alcohol as required by the study restrictions (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of spirits)
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic

For participants with T2DM :

* Have had heart disease or stroke within 6 months before entering the study
* Have health complications due to poorly controlled diabetes as shown by blood and urine laboratory test results or based on physical examination and medical assessment as determined by the study doctor
* Have been hospitalized for poor control of diabetes (keto-acidotic episode) in the last 6 months
* Have used insulin to control diabetes in the last 1 year
* Show symptoms of high blood sugar (for example, frequent urination, always feeling thirsty, or unexpected weight loss)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 ) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single ascending dose crossover study with 2 parts and 3 periods per part. Part A had 3 cohorts (healthy participants). Part B had 1 cohort [with type 2 diabetes mellitus (T2DM)]. Participants in Part A, Cohort 3 completed 2 periods, as ninth (contingency) dose not tested based on interim data. There was ≥10 days between dosing for any participant.
Groups:
- Part A, Cohort 1, Sequence 1: Healthy participants received a single oral dose of the following:
  Period 1: Placebo
  Period 2: 1.5 milligrams (mg) LY2922083
  Period 3: 5 mg LY2922083
- Part A, Cohort 1, Sequence 2: Healthy participants received a single oral dose of the following:
  Period 1: 0.5 mg LY2922083
  Period 2: Placebo
  Period 3: 5 mg LY2922083
- Part A, Cohort 1, Sequence 3: Healthy participants received a single oral dose of the following:
  Period 1: 0.5 mg LY2922083
  Period 2: 1.5 mg LY2922083
  Period 3: Placebo
- Part A, Cohort 2, Sequence 1: Healthy participants received a single oral dose of the following:
  Period 1: Placebo
  Period 2: 50 mg LY2922083
  Period 3: 150 mg LY2922083
- Part A, Cohort 2, Sequence 2: Healthy participants received a single oral dose of the following:
  Period 1: 15 mg LY2922083
  Period 2: Placebo
  Period 3: 150 mg LY2922083
- Part A, Cohort 2, Sequence 3: Healthy participants received a single oral dose of the following:
  Period 1: 15 mg LY2922083
  Period 2: 50 mg LY2922083
  Period 3: Placebo
- Part A, Cohort 3, Sequence 1: Healthy participants received a single oral dose of the following:
  Period 1: Placebo
  Period 2: 845 mg LY2922083
- Part A, Cohort 3, Sequence 2: Healthy participants received a single oral dose of the following:
  Period 1: 450 mg LY2922083
  Period 2: Placebo
- Part A, Cohort 3, Sequence 3: Healthy participants received a single oral dose of the following:
  Period 1: 450 mg LY2922083
  Period 2: 845 mg LY2922083
- Part B, Cohort 1, Sequence 1: Participants with T2DM received a single oral dose of the following:
  Period 1: Placebo
  Period 2: 450 mg LY2922083
  Period 3: 845 mg LY2922083
- Part B, Cohort 1, Sequence 2: Participants with T2DM received a single oral dose of the following:
  Period 1: 150 mg LY2922083
  Period 2: Placebo
  Period 3: 845 mg LY2922083
- Part B, Cohort 1, Sequence 3: Participants with T2DM received a single oral dose of the following:
  Period 1: 150 mg LY2922083
  Period 2: 450 mg LY2922083
  Period 3: Placebo
Period: Intervention Period 1 and Washout
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 1 | Part A, Cohort 2, Sequence 2 | Part A, Cohort 2, Sequence 3 | Part A, Cohort 3, Sequence 1 | Part A, Cohort 3, Sequence 2 | Part A, Cohort 3, Sequence 3 | Part B, Cohort 1, Sequence 1 | Part B, Cohort 1, Sequence 2 | Part B, Cohort 1, Sequence 3
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2 and Washout
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 1 | Part A, Cohort 2, Sequence 2 | Part A, Cohort 2, Sequence 3 | Part A, Cohort 3, Sequence 1 | Part A, Cohort 3, Sequence 2 | Part A, Cohort 3, Sequence 3 | Part B, Cohort 1, Sequence 1 | Part B, Cohort 1, Sequence 2 | Part B, Cohort 1, Sequence 3
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Contingency dose not tested | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 0 | 0
Period: Intervention Period 3 and Washout
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 1 | Part A, Cohort 2, Sequence 2 | Part A, Cohort 2, Sequence 3 | Part A, Cohort 3, Sequence 1 | Part A, Cohort 3, Sequence 2 | Part A, Cohort 3, Sequence 3 | Part B, Cohort 1, Sequence 1 | Part B, Cohort 1, Sequence 2 | Part B, Cohort 1, Sequence 3
Started | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study drug or placebo, and had at least 1 postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Cohort 1, Sequence 1 | Part A, Cohort 1, Sequence 2 | Part A, Cohort 1, Sequence 3 | Part A, Cohort 2, Sequence 1 | Part A, Cohort 2, Sequence 2 | Part A, Cohort 2, Sequence 3 | Part A, Cohort 3, Sequence 1 | Part A, Cohort 3, Sequence 2 | Part A, Cohort 3, Sequence 3 | Part B, Cohort 1, Sequence 1 | Part B, Cohort 1, Sequence 2 | Part B, Cohort 1, Sequence 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 3 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Serious Adverse Event(s) (SAEs)
Description: Events deemed by the Investigator to be SAEs related to study drug administration are reported. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion (up to 70 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Parts A and B): Healthy participants or participants with T2DM, in Part A or B, Cohorts 1, 2, or 3, who received a single oral dose of placebo in 1 of 3 study periods.
- 0.5 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 1 who received a single oral dose of 0.5 mg LY2922083 in study period 1.
- 1.5 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 1 who received a single oral dose of 1.5 mg LY2922083 in study period 2.
- 5 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 1 who received a single oral dose of 5 mg LY2922083 in study period 3.
- 15 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 2 who received a single oral dose of 15 mg LY2922083 in study period 1.
- 50 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 2 who received a single oral dose of 50 mg LY2922083 in study period 2.
- 150 mg LY2922083 (Parts A and B): Healthy participants in Part A, Cohort 2 who received a single oral dose of 150 mg LY2922083 in study period 3 and participants with T2DM in Part B, Cohort 1 who received a single oral dose of 150 mg LY2922083 in study period 1.
- 450 mg LY2922083 (Parts A and B): Healthy participants in Part A, Cohort 3 who received a single oral dose of 450 mg LY2922083 in study period 1 and participants with T2DM in Part B, Cohort 1 who received a single oral dose of 450 mg LY2922083 in study period 2.
- 845 mg LY2922083 (Parts A and B): Healthy participants in Part A, Cohort 3 who received a single oral dose of 845 mg LY2922083 in study period 2 and participants with T2DM in Part B, Cohort 1 who received a single oral dose of 845 mg LY2922083 in study period 3.
Arm/Group | Placebo (Parts A and B) | 0.5 mg LY2922083 (Part A) | 1.5 mg LY2922083 (Part A) | 5 mg LY2922083 (Part A) | 15 mg LY2922083 (Part A) | 50 mg LY2922083 (Part A) | 150 mg LY2922083 (Parts A and B) | 450 mg LY2922083 (Parts A and B) | 845 mg LY2922083 (Parts A and B)
Number analyzed (Participants) | 32 | 6 | 6 | 6 | 6 | 6 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve From Time 0 to Infinite Time [AUC(0-∞)] of LY2922083
Time Frame: Predose up to 72 hours (h) after each dose of study drug (Part A: predose, 0.5, 1.5, 2.5, 4, 6, 12, 18, 24, 36, 48 and 72 h postdose. Part B: predose, 0.5, 1.5, 4, 6, 12, 18, 24, 36, 48 and 72 h postdose.)
Population: All participants who received at least 1 dose of the study drug and had sufficient PK data to calculate AUC(0-∞).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Groups:
- 150 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 2 who received a single oral dose of 150 mg LY2922083 in study period 3.
- 450 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 3 who received a single oral dose of 450 mg LY2922083 in study period 1.
- 845 mg LY2922083 (Part A): Healthy participants in Part A, Cohort 3 who received a single oral dose of 845 mg LY2922083 in study period 2.
- 150 mg LY2922083 (Part B): Participants with T2DM in Part B, Cohort 1 who received a single oral dose of 150 mg LY2922083 in study period 1.
- 450 mg LY2922083 (Part B): Participants with T2DM in Part B, Cohort 1 who received a single oral dose of 450 mg LY2922083 in study period 2.
- 845 mg LY2922083 (Part B): Participants with T2DM in Part B, Cohort 1 who received a single oral dose of 845 mg LY2922083 in study period 3.
Arm/Group | 0.5 mg LY2922083 (Part A) | 1.5 mg LY2922083 (Part A) | 5 mg LY2922083 (Part A) | 15 mg LY2922083 (Part A) | 50 mg LY2922083 (Part A) | 150 mg LY2922083 (Part A) | 450 mg LY2922083 (Part A) | 845 mg LY2922083 (Part A) | 150 mg LY2922083 (Part B) | 450 mg LY2922083 (Part B) | 845 mg LY2922083 (Part B)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanograms*hour per milliliter (ng*hr/mL) | 25.9 (38) | 79.5 (47) | 220 (52) | 612 (25) | 1560 (28) | 3270 (34) | 10200 (23) | 16900 (42) | 4900 (117) | 10400 (60) | 24400 (89)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY2922083
Time Frame: Predose up to 72 h after each dose of study drug (Part A: predose, 0.5, 1.5, 2.5, 4, 6, 12, 18, 24, 36, 48 and 72 h postdose. Part B: predose, 0.5, 1.5, 4, 6, 12, 18, 24, 36, 48 and 72 h postdose.)
Population: All participants who received at least 1 dose of the study drug and had sufficient PK data to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.5 mg LY2922083 (Part A) | 1.5 mg LY2922083 (Part A) | 5 mg LY2922083 (Part A) | 15 mg LY2922083 (Part A) | 50 mg LY2922083 (Part A) | 150 mg LY2922083 (Part A) | 450 mg LY2922083 (Part A) | 845 mg LY2922083 (Part A) | 150 mg LY2922083 (Part B) | 450 mg LY2922083 (Part B) | 845 mg LY2922083 (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 2.36 (48) | 8.64 (25) | 20.3 (29) | 66.0 (41) | 152 (18) | 327 (67) | 927 (49) | 1720 (44) | 407 (131) | 808 (50) | 2220 (73)

4. Secondary Outcome: Change From Baseline in Blood Glucose Area Under the Effective Concentration Curve From Time 0 to 24 h Postdose [AUEC(0-24)]
Description: Least Squares (LS) mean values were adjusted for baseline, treatment, period, treatment sequence, participant and error.
Time Frame: Baseline (predose for Part A and Day -1 time-matched for Part B), up to 24 h postdose (1.5, 2.5, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 18, and 24 h postdose)
Population: All participants who received at least 1 dose of the study drug or placebo and had sufficient pharmacodynamic data to calculate glucose AUEC(0-24).
Measure: Least Squares Mean (Standard Error); unit: millimoles*hour per liter (mmol*h/L)
Groups:
- Placebo (Part A): Healthy participants in Part A, Cohorts 1, 2, or 3 who received a single oral dose of placebo in 1 of 3 study periods.
- Placebo (Part B): Participants with T2DM in Part B, Cohort 1 who received a single oral dose of placebo in 1 of 3 study periods.
Arm/Group | Placebo (Part A) | 0.5 mg LY2922083 (Part A) | 1.5 mg LY2922083 (Part A) | 5 mg LY2922083 (Part A) | 15 mg LY2922083 (Part A) | 50 mg LY2922083 (Part A) | 150 mg LY2922083 (Part A) | 450 mg LY2922083 (Part A) | 845 mg LY2922083 (Part A) | Placebo (Part B) | 150 mg LY2922083 (Part B) | 450 mg LY2922083 (Part B) | 845 mg LY2922083 (Part B)
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
millimoles*hour per liter (mmol*h/L) | 7.08 (1.17) [NA to NA] | 6.32 (2.86) [-5.40 to 3.90] | -0.02 (2.84) [-11.70 to -2.49] | 12.34 (2.78) [0.20 to 10.34] | 8.88 (3.00) [-2.93 to 6.55] | 8.40 (2.94) [-3.32 to 5.98] | 4.78 (2.73) [-7.24 to 2.65] | 6.13 (2.87) [-6.00 to 4.11] | 3.68 (2.87) [-8.45 to 1.65] | 4.60 (1.90) [NA to NA] | 8.48 (3.56) [7.92 to 24.85] | 1.18 (3.18) [-26.99 to 10.89] | 3.05 (3.24) [-26.92 to -12.05]

5. Secondary Outcome: Change From Baseline in C-Peptide Area Under the Effective Concentration Curve From Time 0 to 6 h Postdose [AUEC(0-6)]
Description: LS mean values were adjusted for baseline, treatment, period, treatment sequence, participant and error.
Time Frame: Baseline (predose for Part A and Day -1 time-matched for Part B), up to 6 h postdose (1.5, 2.5, 4, 4.5, 5, and 6 h postdose)
Population: All participants who received at least 1 dose of the study drug or placebo and had sufficient pharmacodynamic data to calculate C-peptide AUEC(0-6).
Measure: Least Squares Mean (Standard Error); unit: picomoles*hour per liter (pmol*h/L)
Groups:
- Placebo (Part B): Participants with T2DM in Part B, Cohorts 1, 2, or 3 who received a single oral dose of placebo in 1 of 3 study periods.
Arm/Group | Placebo (Part A) | 0.5 mg LY2922083 (Part A) | 1.5 mg LY2922083 (Part A) | 5 mg LY2922083 (Part A) | 15 mg LY2922083 (Part A) | 50 mg LY2922083 (Part A) | 150 mg LY2922083 (Part A) | 450 mg LY2922083 (Part A) | 845 mg LY2922083 (Part A) | Placebo (Part B) | 150 mg LY2922083 (Part B) | 450 mg LY2922083 (Part B) | 845 mg LY2922083 (Part B)
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
picomoles*hour per liter (pmol*h/L) | 6638.85 (557.21) | 6518.87 (1195.43) | 8107.68 (1194.99) | 5742.81 (1172.87) | 8283.17 (1225.04) | 6715.88 (1221.10) | 5653.51 (1140.26) | 4525.49 (1204.61) | 5554.47 (1203.47) | 1670.60 (580.54) | 2865.28 (1174.05) | 1061.59 (1178.54) | 512.14 (1180.77)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to 70 days)
Arm/Group | Placebo (Parts A and B) | 0.5 mg LY2922083 (Part A) | 1.5 mg LY2922083 (Part A) | 5 mg LY2922083 (Part A) | 15 mg LY2922083 (Part A) | 50 mg LY2922083 (Part A) | 150 mg LY2922083 (Parts A and B) | 450 mg LY2922083 (Parts A and B) | 845 mg LY2922083 (Parts A and B)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/32 | 1/6 | 2/6 | 0/6 | 2/6 | 5/6 | 9/12 | 8/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Parts A and B) (N=32) | 0.5 mg LY2922083 (Part A) (N=6) | 1.5 mg LY2922083 (Part A) (N=6) | 5 mg LY2922083 (Part A) (N=6) | 15 mg LY2922083 (Part A) (N=6) | 50 mg LY2922083 (Part A) (N=6) | 150 mg LY2922083 (Parts A and B) (N=12) | 450 mg LY2922083 (Parts A and B) (N=12) | 845 mg LY2922083 (Parts A and B) (N=12)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 3 (4)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes